CLINICAL TRIAL: NCT07131306
Title: National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM): To Study the Safety and Efficacy of Mesenchymal Stem-Cell (MSC) Therapy in the Management of Non-viral ACLF Patients: Phase-II Clinical Study
Brief Title: National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM): Evaluating Mesenchymal Stem Cell Therapy in Non-viral Acute on Chronic Liver Failure (ACLF) Patient- Phase-II Trial
Acronym: NC-CHRM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-71
Record Dates: First submitted 2025-07-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute on Chronic Liver Failure; Mesenchymal Stem Cells; ACLF; Liver Regeneration
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord mesenchymal stem cell (ucMSC) and Standard medical treatment (SMT) (Experimental): Patient randomize for MSC therapy together with standard medical treatment, ucMSC 1 million/kg will be given once a week for 4 week . 250 ml normal saline will be infused 30 minutes prior to ucMSCs infusion. The fresh ucMSCs will then be infused through IV canula peripherally over 30 minutes followed by a further 250 ml normal saline over 20-30 minutes. A baseline early warning score (EWS) will be undertaken with continuous monitoring of pulse and with blood pressure checks every 5 minutes during the cell infusion and then every 15 minutes during the subsequent 2-hour observation period, then every hour for the remaining 10-hour observation period (minimum total of 12 hours observation) after cell infusion. All patients will receive the standard medical treatment.
  Interventions: Drug: ucMSC and Standard medical treatment; Other: Standard medical treatment
- Standard Medical Treatment (Active Comparator): Patients in the SMT group will be managed as per requirement with nutrition, lactulose, intravenous albumin, fluids, blood transfusion or antibiotics as required. Patients with hepatorenal syndrome will be treated with intravenous terlipressin or noradrenaline. Renal replacement therapy will be done for standard indications in patients with severe volume overload, metabolic acidosis, or hyperkalemia unresponsive to goal-directed SMT as described above. Mechanical ventilation and routine intensive care management will be done in patients with multiorgan failure.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: ucMSC and Standard medical treatment — umbilical cord Mesenchymal stem cell1 million/kg will be given once a week for 4 week . 250 ml normal saline will be infused 30 minutes prior to ucMSCs infusion. All patients will receive the standard medical treatment.
  Arms: Umbilical cord mesenchymal stem cell (ucMSC) and Standard medical treatment (SMT)
Other: Standard medical treatment — Standard medical treatment

SUMMARY:
Liver disease deaths are rising, but transplants remain scarce in India. With over 100,000 needed annually and only ~2,500 performed, non-transplant options are urgently needed. Regenerative therapy, especially MSCs, shows promise but lacks validation, particularly for non-viral ACLF. The proposed NC-CHRM aims to develop and validate MSC-based therapy to promote native liver regeneration and offer a safe, effective, transplant-free treatment.

DETAILED DESCRIPTION:
The incidence of deaths from chronic liver diseases (CLD) and cirrhosis are rapidly increasing globally, including India. Liver transplant is the only curative option. Unfortunately, transplant is often not feasible. There is a need for nearly 100,000 liver transplants every year in India, though, only about 2,500 transplants are being done at present across the country. There is therefore, a huge unmet need of developing non-transplant options for chronic liver disease patients. In this regard emerging science of regenerative therapy holds great promises but therapeutic benefit of these therapies is limited due to lack of clinical validation.

Novelty: Liver failure is failure of regeneration hence, potentiating native liver repair and regeneration can serve as potential non-transplant approaches. Others and us have shown in experimental studies that mesenchymal stem cells (MSCs) can improve hepatic regeneration. MSC therapy trials in decompensated cirrhosis and viral ACLF in Korea, China and Japan have shown promise but their utility in non-viral ACLF is limited. In the proposed National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM) we will use this novel regenerative medicine approaches MSC for management of acute liver failure in non-viral ACLF to develop safe and effective regenerative therapy clinical protocol for transplant free management of liver failure in cirrhosis. Using integrated cellular, molecular and functional analysis we will also establish their mechanism of action and identify biomarker to access therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* ACLF patients with Model for End-Stage Liver Disease(MELD)>18 or APASL ACLF Research Consortium(AARC) grade 2 or more with (no or single extrahepatic organ dysfunction or failure having no option of liver transplant).

Exclusion Criteria:

* Age <18 or >65 yrs
* Patients with active sepsis
* Patients with hepatic venous outflow tract obstruction (HVOTO) or Extrahepatic portal vein obstruction (EHPVO)
* Hepatocellular carcinoma (beyond Milan) or any extrahepatic malignancy
* Active bleed (mucosal or variceal) or severe coagulopathy (platelets <20,000 or INR>4)
* Patients with refractory shock requiring norepinephrine >0.5ug/kg/min
* Patients with severe Acute Respiratory Distress Syndrome (ARDS) with Pa02/Fi02 <150
* Patients with retroviral infections
* Autoimmune hepatitis
* Viral etiology of liver disease
* Co-existent Hepatitis B, Hepatitis C, HIV
* Chronic kidney disease
* Multiorgan failure or Disseminated Intravascular Coagulation (DIC)
* Patients improving on standard medical treatment
* Patients on immunosuppressive medications
* Pregnancy or active breastfeeding
* Known severe cardiopulmonary diseases (structural or valvular heart disease, coronary artery disease, coronary pulmonary disease, chronic kidney disease)
* Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
90-day transplant-free survival | 90-day

SECONDARY OUTCOMES:
28-day and 6-month transplant free survival | 28-day and 6-month
Cumulative incidence of AKI, sepsis and extrahepatic-extrarenal organ dysfunctions at day 28, day 60 and day 90. | Day 28, day 60 and day 90.
Proportion of patients achieving resolution of ACLF (complete and partial) at day 90. | Day 90
Improvement in liver severity indices MELD score by 4 points and improvement in AARC grade by 1 from baseline at 28 days, day 60 and day 90. | Day 28, Day 60 and Day 90.
Impact on liver injury and regeneration (serum and histology ) at day 28 and day 90. | Day 28 and day 90
Change in monocyte energy metabolism (glycolysis and OXPHOS test) and function from baseline at day 3, day 7, day 28 and day 90. | Day 3, 7,28 and 90
Change in peripheral blood level of cytokines (pro-inflammatory: TNF-α, IL-6, IL-1β; anti-inflammatory: IL-10, TGF-β), endotoxin and extracellular vesicles (EVs, number of EVs per mL of blood) at baseline, day 3, day14, day 28 and day 90. | Day 3,14, 28, 90
Proportion of patients completing treatment without major adverse effects | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided